CLINICAL TRIAL: NCT04018417
Title: A Randomized, Double-masked, Placebo-controlled Study of the Safety of Amphotericin 0.255 μg/mL in Optisol-GS
Brief Title: Evaluation of Amphotericin B in Optisol-GS for Prevention of Post-Keratoplasty Fungal Infections.
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Reconsidered significance in light of newly published in vitro data.
Sponsor: Cornea Research Foundation of America (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2019-005
Record Dates: First submitted 2019-07-11; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Fuchs' Endothelial Dystrophy
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy | interventions — Amphotericin B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Amphotericin B (Experimental): The eye bank will add amphotericin B 0.255 μg/mL to the Optisol-GS donor cornea storage solution.
  Interventions: Drug: Amphotericin B
- Control (No Intervention): The donor cornea will be stored in Optisol-GS per the eye bank's standard procedure.

INTERVENTIONS:
Drug: Amphotericin B — Drug concentration: 0.255 μg/mL
  Arms: Amphotericin B

SUMMARY:
With the increasing popularity of endothelial keratoplasty, a coincident increase in the rate of fungal infections post-keratoplasty has been seen in the United States. In this study, the eye bank will harvest pairs of donor corneas and randomize one cornea from each pair to be stored in Optisol-GS per Eye Bank Association of America guidelines. The eye bank will add amphotericin B 0.255 μg/mL (antifungal) to the storage solution for the mate cornea. The study donor corneas will be assigned to participants who are scheduled to undergo Descemet membrane endothelial keratoplasty. The surgeons, participants, and evaluators will remain masked regarding the donor cornea storage solution assignment. The participants will be followed for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female at least 18 years of age and any race or ethnicity
* Scheduled to have Descemet membrane endothelial keratoplasty

Exclusion Criteria:

* History of glaucoma surgery in operative eye
* Known allergy or intolerance to amphotericin B
* Presence of anterior chamber intraocular lens
* Corneal stromal or epithelial dysfunction
* Presence of glaucoma defined as optic nerve damage as confirmed on Humphrey visual field testing or retinal nerve fiber layer analysis
* Presence of peripheral anterior synechiae

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2019-07-03 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
Endothelial cell density | 6 months
  Central corneal endothelial cell density will be assessed by specular microscopy

SECONDARY OUTCOMES:
Incidence of post-keratoplasty fungal keratitis | 6 months
  The incidence of post-keratoplasty fungal keratitis will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr, MD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Aldave AJ, DeMatteo J, Glasser DB, Tu EY, Iliakis B, Nordlund ML, Misko J, Verdier DD, Yu F. Report of the Eye Bank Association of America medical advisory board subcommittee on fungal infection after corneal transplantation. Cornea. 2013 Feb;32(2):149-54. doi: 10.1097/ICO.0b013e31825e83bf. PMID 23051906
- [Background] Armitage WJ. Preservation of Human Cornea. Transfus Med Hemother. 2011;38(2):143-147. doi: 10.1159/000326632. Epub 2011 Mar 16. PMID 21566714
- [Background] Hassan SS, Wilhelmus KR; Medical Review Subcommittee of the Eye Bank Association of America. Eye-banking risk factors for fungal endophthalmitis compared with bacterial endophthalmitis after corneal transplantation. Am J Ophthalmol. 2005 Apr;139(4):685-90. doi: 10.1016/j.ajo.2004.12.016. PMID 15808165
- [Background] Hassan SS, Wilhelmus KR, Dahl P, Davis GC, Roberts RT, Ross KW, Varnum BH; Medical Review Subcommittee of the Eye Bank Association of America. Infectious disease risk factors of corneal graft donors. Arch Ophthalmol. 2008 Feb;126(2):235-9. doi: 10.1001/archophthalmol.2007.45. PMID 18268215
- [Background] Keyhani K, Seedor JA, Shah MK, Terraciano AJ, Ritterband DC. The incidence of fungal keratitis and endophthalmitis following penetrating keratoplasty. Cornea. 2005 Apr;24(3):288-91. doi: 10.1097/01.ico..0000138832.3486.70. PMID 15778600
- [Background] Merchant A, Zacks CM, Wilhelmus K, Durand M, Dohlman CH. Candidal endophthalmitis after keratoplasty. Cornea. 2001 Mar;20(2):226-9. doi: 10.1097/00003226-200103000-00026. PMID 11248837
- [Background] Doshi H, Pabon S, Price MO, Feng MT, Price FW Jr. Overview of Systemic Candida Infections in Hospital Settings and Report of Candida After DMEK Successfully Treated With Antifungals and Partial Graft Excision. Cornea. 2018 Aug;37(8):1071-1074. doi: 10.1097/ICO.0000000000001608. PMID 29634675
- [Background] Duncan K, Parker J, Hoover C, Jeng BH. The Effect of Light Exposure on the Efficacy and Safety of Amphotericin B in Corneal Storage Media. JAMA Ophthalmol. 2016 Apr;134(4):432-6. doi: 10.1001/jamaophthalmol.2016.0008. PMID 26914028
- [Background] Lopez RM, Ayestaran A, Pou L, Montoro JB, Hernandez M, Caragol I. Stability of amphotericin B in an extemporaneously prepared i.v. fat emulsion. Am J Health Syst Pharm. 1996 Nov 15;53(22):2724-7. doi: 10.1093/ajhp/53.22.2724. PMID 8931814